CLINICAL TRIAL: NCT02709538
Title: A Double-Blind, Randomized, Parallel-Group Study to Evaluate Long-Term Safety, Tolerability, and Efficacy of a Fixed Dose Combination GSP 301 Nasal Spray Compared With Two Placebo Nasal Spray Formulations in Subjects (Aged 12 Years and Older) With Perennial Allergic Rhinitis (PAR)
Brief Title: Long Term Safety and Efficacy of Fixed Dose Combination GSP 301 Nasal Spray (NS) in the Treatment of Perennial Allergic Rhinitis (PAR)
Acronym: GSP 301-303
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glenmark Specialty S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GPL/CT/2014/018/III
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- GSP 301 NS (Experimental)
  Interventions: Drug: GSP 301 NS
- GSP 301 Placebo NS pH 3.7 (Placebo Comparator)
  Interventions: Drug: GSP 301 Placebo NS pH 3.7
- GSP 301 Placebo NS pH 7.0 (Placebo Comparator)
  Interventions: Drug: GSP 301 Placebo NS pH 7.0

INTERVENTIONS:
Drug: GSP 301 NS — FDC of olopatadine HCl and mometasone furoate: 2 spray in each nostril twice daily for 52 weeks
  Arms: GSP 301 NS
Drug: GSP 301 Placebo NS pH 3.7 — 2 spray in each nostril twice daily for 52 weeks
  Arms: GSP 301 Placebo NS pH 3.7
Drug: GSP 301 Placebo NS pH 7.0 — 2 spray in each nostril twice daily for 52 weeks
  Arms: GSP 301 Placebo NS pH 7.0

SUMMARY:
To evaluate the long term safety and efficacy of GSP 301 NS compared to 2 placebo NS formulations for the treatment of perennial allergic rhinitis (subjects 12 years of age and older)

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥12 years and older inclusive of either sex.
2. Documented clinical history of PAR (for at least 2 years preceding the Screening Visit [Visit 1]) and exhibiting a documented positive skin prick test (wheal diameter at least 3 mm greater than negative diluent control wheal) to at least 1 allergen known to induce PAR. Documentation of a positive result within 12 months prior to the Screening Visit (Visit 1) is acceptable.

Exclusion Criteria:

1. Pregnant or lactating women.
2. History of anaphylaxis and/or other severe local reaction(s) to skin testing.
3. History of positive test for HIV, Hepatitis B or Hepatitis C infection.
4. Documented evidence of acute or significant chronic sinusitis or chronic purulent postnasal drip.
5. Subjects with an active pulmonary disorder or infection.
6. Subjects with posterior subcapsular cataracts or glaucoma

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2016-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh Tantry, Study Director — Glenmark Pharmaceuticals
Locations (34):
- United States (34):
  - Investigational Site 2, Hot Springs, Arkansas
  - Investigational Site 28, Encinitas, California
  - Investigational Site 27, San Diego, California
  - Investigational Site 29, San Diego, California
  - Investigational Site 32, Denver, Colorado
  - Investigational Site 26, Aventura, Florida
  - Investigational Site 9, Miami, Florida
  - Investigational Site 33, Tallahassee, Florida
  - Investigational Site 11, Stockbridge, Georgia
  - Investigational Site 4, Louisville, Kentucky
  - Investigational Site 5, Bethesda, Maryland
  - Investigational Site 15, St Louis, Missouri
  - Investigational Site 30, Bellevue, Nebraska
  - Investigational Site 19, Skillman, New Jersey
  - Investigational Site 18, Corning, New York
  - Investigational Site 7, High Point, North Carolina
  - Investigational Site 21, Raleigh, North Carolina
  - Investigational Site 16, Sylvania, Ohio
  - Investigational Site 22, Pittsburgh, Pennsylvania
  - Investigational Site 13, Spartanburg, South Carolina
  - Investigational Site 23, Austin, Texas
  - Investigational Site 24, Austin, Texas
  - Investigational Site 3, Austin, Texas
  - Investigational Site 31, Dallas, Texas
  - Investigational Site 34, El Paso, Texas
  - Investigational Site 6, Kerrville, Texas
  - Investigational Site 14, New Braunfels, Texas
  - Investigational Site 10, San Antonio, Texas
  - Investigational Site 12, San Antonio, Texas
  - Investigational Site 17, San Antonio, Texas
  - Investigational Site 1, San Antonio, Texas
  - Investigational Site 20, San Antonio, Texas
  - Investigational Site 25, Waco, Texas
  - Investigational Site 8, Waco, Texas

REFERENCES:
- [Derived] Segall N, Prenner B, Lumry W, Caracta CF, Tantry SK. Long-term safety and efficacy of olopatadine-mometasone combination nasal spray in patients with perennial allergic rhinitis. Allergy Asthma Proc. 2019 Sep 1;40(5):301-310. doi: 10.2500/aap.2019.40.4233. Epub 2019 Jun 27. PMID 31248471

RESULTS

PARTICIPANT FLOW:
Groups:
- GSP 301 NS: GSP 301 NS: 2 spray in each nostril twice daily for 52 weeks
Period: Overall Study
Arm/Group | GSP 301 NS | GSP 301 Placebo NS pH 3.7 | GSP 301 Placebo NS pH 7.0
Started | 400 | 100 | 101
Completed | 287 | 72 | 81
Not Completed | 113 | 28 | 20
Not completed — Adverse Event | 13 | 2 | 3
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 24 | 8 | 4
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 40 | 7 | 4
Not completed — Non-compliance with study procedures | 5 | 0 | 0
Not completed — Non-compliance with study drug | 2 | 0 | 0
Not completed — Protocol deviation | 10 | 4 | 4
Not completed — Withdrawal by Parent or Legal Guardian | 1 | 0 | 0
Not completed — Other | 16 | 7 | 5

BASELINE CHARACTERISTICS:
Population: Participants at the baseline measurement are less than that started because some subjects were not randomized or did not use the study drug on at least one occasion.
Groups:
- Total: Total of all reporting groups
Arm/Group | GSP 301 NS | GSP 301 Placebo NS pH 3.7 | GSP 301 Placebo NS pH 7.0 | Total
Number analyzed (Participants) | 393 | 99 | 101 | 593
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (14.8) | 42.1 (15.4) | 41.2 (13.5) | 40.8 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 269 | 68 | 68 | 405
  Male | 124 | 31 | 33 | 188
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 10 | 1 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 95 | 17 | 22 | 134
  White | 282 | 78 | 76 | 436
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs).
Description: All TEAEs and serious adverse events (SAEs) occurring in the study, in terms of nature, onset, duration, severity, relationship, and outcome were reported.
Time Frame: 52 weeks
Population: Safety Analysis Set (SAS) will consist of all subjects who took at least 1 dose of study medication following randomization. This was the primary analysis set for safety analyses.
Measure: Number; unit: participants
Arm/Group | GSP 301 NS | GSP 301 Placebo NS pH 3.7 | GSP 301 Placebo NS pH 7.0
Number analyzed (Participants) | 393 | 99 | 101
participants | 203 | 41 | 54

ADVERSE EVENTS:
Time Frame: The AEs and SAEs were collected from the time of signing the informed consent form until the end of study until 52 weeks.
Description: Total number of Participants at Risk is consistent with the number of participants reported at Baseline measurement. These participant numbers are not consistent with the numbers provided in the Participant Flow module because some of the subjects from the 'Total number at the start' were not randomized in the study or did not use the study drug on at least one occasion.
Arm/Group | GSP 301 NS | GSP 301 Placebo NS pH 3.7 | GSP 301 Placebo NS pH 7.0
All-Cause Mortality (participants affected / at risk) | 0/393 | 0/99 | 0/101
Serious Adverse Events (participants affected / at risk) | 7/393 | 2/99 | 2/101
Other Adverse Events (participants affected / at risk) | 72/393 | 15/99 | 25/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSP 301 NS (N=393) | GSP 301 Placebo NS pH 3.7 (N=99) | GSP 301 Placebo NS pH 7.0 (N=101)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSP 301 NS (N=393) | GSP 301 Placebo NS pH 3.7 (N=99) | GSP 301 Placebo NS pH 7.0 (N=101)
Nasopharyngitis (Infections and infestations) | 12 (14) | 5 (6) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 25 (30) | 6 (8) | 9 (12)
Headache (Nervous system disorders) | 16 (18) | 3 (3) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (23) | 2 (2) | 2 (3)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 11 (15) | 2 (2) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/38/NCT02709538/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT02709538/SAP_001.pdf